CLINICAL TRIAL: NCT07401173
Title: A Prospective, Multicenter, Observational Study Validating the Multimodal Deep Learning Radiomics Model (DeepComp) for Preoperative Prediction of Major Postoperative Complications in Patients With Gastric Cancer
Brief Title: DeepComp for Prediction of Gastric Cancer Postoperative Complications (DeepComp-Prospective)
Status: Not yet recruiting | Type: Observational
Sponsor: Qun Zhao (Other)
Responsible Party: Sponsor-Investigator, Qun Zhao, Professor, Hebei Medical University
Organization: Hebei Medical University (Other)
Other Study IDs: DeepComp-Pro-001
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Gastric Cancer (Diagnosis); Postoperative Complications
MeSH Terms: conditions — Stomach Neoplasms; Disease; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days

GROUPS / COHORTS (1):
- Gastric Cancer Surgery Cohort: Patients diagnosed with gastric cancer who are scheduled to undergo radical gastrectomy (open, laparoscopic, or robotic). All participants will receive standard preoperative contrast-enhanced CT scans. The DeepComp AI model will be applied to these scans to predict the risk of postoperative complications.

SUMMARY:
Gastric cancer is a leading cause of cancer-related mortality, and radical surgery remains the primary treatment. However, postoperative complications are common and can significantly impact patient recovery and quality of life. Currently, doctors lack precise tools to accurately predict which patients are at high risk for developing severe complications before surgery.

This study aims to validate a novel artificial intelligence (AI) model called "DeepComp." The DeepComp model integrates clinical data with advanced radiomic features derived from routine preoperative CT scans. Specifically, it analyzes both the tumor characteristics and the patient's body composition (including skeletal muscle and fat distribution) to assess physiological reserve.

In this prospective, multicenter observational study, researchers will enroll patients scheduled for gastric cancer surgery across five medical centers. The DeepComp model will be used to predict the risk of moderate-to-severe postoperative complications (Clavien-Dindo grade II or higher). These predictions will then be compared with the actual clinical outcomes observed 30 days after surgery. The goal is to determine the accuracy and reliability of the DeepComp model in a real-world clinical setting, potentially providing a powerful tool for personalized surgical risk assessment.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years.

Histologically confirmed gastric adenocarcinoma.

Scheduled for elective radical gastrectomy (open, laparoscopic, or robotic) with curative intent.

Standard preoperative contrast-enhanced abdominal CT scans (venous phase) performed within 14 days prior to surgery.

Willingness to sign informed consent.

Exclusion Criteria:

Emergency surgery due to perforation, obstruction, or massive bleeding.

Intraoperative findings of distant metastasis (Stage IV) or unresectable disease preventing R0 resection.

Concurrent or previous malignant tumors within the last 5 years (except gastric cancer).

Pregnancy or lactation.

Severe metallic artifacts on CT images preventing radiomic analysis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with potentially resectable gastric cancer who are admitted to the participating centers for surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Postoperative Complications (Clavien-Dindo Grade ≥ II) | Postoperative 30 days
  Postoperative complications will be graded according to the Clavien-Dindo classification system. Major complications are defined as Grade II or higher, which require pharmacological treatment, surgical/endoscopic/radiological intervention, or life-threatening complications (including death). The occurrence of these events will be recorded and compared with the model's preoperative predictions.

SECONDARY OUTCOMES:
Predictive Performance of the DeepComp Model (AUC) | Postoperative 30 days
  The discrimination performance of the DeepComp model in predicting major postoperative complications will be evaluated using the Area Under the Receiver Operating Characteristic Curve (AUC). Sensitivity, specificity, positive predictive value, and negative predictive value will also be calculated.
Length of Hospital Stay | Up to 30 days
  Defined as the number of days from surgery to discharge.